CLINICAL TRIAL: NCT03280056
Title: A Phase 3, Randomized Double-Blind, Placebo-Controlled Multicenter Study to Evaluate Efficacy and Safety of Repeated Administration of NurOwn® (Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors) in Participants With ALS
Brief Title: Safety and Efficacy of Repeated Administrations of NurOwn® in ALS Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brainstorm-Cell Therapeutics (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCT-002-US
Record Dates: First submitted 2017-08-29; First posted 2017-09-12 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: MSC; Autologous; Neurotrophic factors
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Multicenter Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind study where the investigators, participants and all sponsor and CRO personnel involved in the conduct, data management or analysis of the study will remain blinded to the treatment assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NurOwn® (MSC-NTF cells) (Active Comparator): Three Intrathecal administrations of NurOwn® (MSC-NTF cells) at bi-monthly intervals
  Interventions: Biological: NurOwn® (MSC-NTF cells); Other: Bone Marrow aspiration
- Placebo (Placebo Comparator): Three Intrathecal administrations of Placebo at bi-monthly intervals
  Interventions: Other: Placebo; Other: Bone Marrow aspiration

INTERVENTIONS:
Biological: NurOwn® (MSC-NTF cells) — NurOwn® (MSC-NTF): One course of treatment that includes three separate intrathecal injections of 100-125 x 10^6 cells every 8 weeks
  NurOwn® (MSC-NTF): Autologous, bone marrow-derived, mesenchymal stem cells secreting neurotrophic factors
  Arms: NurOwn® (MSC-NTF cells)
Other: Placebo — One course of treatment that includes three separate intrathecal injections of Placebo every 8 weeks
  Placebo: liquid solution in syringe for injection
  Arms: Placebo
Other: Bone Marrow aspiration — Bone Marrow aspiration

SUMMARY:
This study will evaluate the safety and efficacy of repeated administration of NurOwn® (MSC-NTF cells) therapy, which is based on transplantation of autologous bone marrow derived mesenchymal stromal cells (MSC), which are enriched from the patient's own bone marrow, propagated ex vivo and induced to secrete Neurotrophic factors (NTFs).

The autologous NurOwn® (MSC-NTF cells) are back-transplanted into the patient intrathecally by standard lumbar puncture where neurons and glial cells are expected to take up the neurotrophic factors secreted by the transplanted cells

DETAILED DESCRIPTION:
Neurotrophic factors (NTFs) are potent survival factors for embryonic, neonatal, and adult neurons and are considered potential therapeutic candidates for ALS. Delivery of multiple NTFs to the immediate environment of afflicted neurons in ALS patients is expected to improve their survival and thus slow down disease progression and alleviate symptoms. NTF-secreting mesenchymal stromal cells (MSC-NTF cells) are a novel cell-therapeutic approach aimed at effectively delivering NTFs directly to the site of damage in ALS patients.

Participants meeting the inclusion and exclusion criteria will be randomized and will undergo bone-marrow aspiration. MSC of the participants randomized to the treatment group will be induced into MSC-NTF cells. Participants will undergo a total of three intrathecal (IT) transplantations with NurOwn® (MSC-NTF cells) or matching placebo at three bi-monthly intervals

ELIGIBILITY:
Inclusion Criteria:

* ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria.
* Having onset of ALS disease symptoms, including limb weakness within 24 months at the Screening Visit.
* ALSFRS-R ≥ 25 at the screening Visit.
* Upright slow vital capacity (SVC) measure ≥ 65% of predicted for gender, height, and age at the screening Visit.
* Rapid progressors
* Participants taking a stable dose of Riluzole are permitted in the study
* Citizen or permanent resident of the United States or Canadian citizen able to travel to a US site for all follow-up study visits

Exclusion Criteria:

* Prior stem cell therapy of any kind
* History of autoimmune or other serious disease (including malignancy and immune deficiency) that may confound study results
* Current use of immunosuppressant medication or anticoagulants (per Investigator discretion)
* Exposure to any other experimental agent or participation in an ALS clinical trial within 30 days prior to Screening Visit
* Use of RADICAVA (edaravone injection) within 30 days of screening or intent to use edaravone at any time during the course of the study including the follow up period
* Use of non-invasive ventilation (BIPAP), diaphragm pacing system or invasive ventilation (tracheostomy)
* Feeding tube
* Pregnant women or women currently breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 196 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit E. Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital; Robert H. Brown, MD, PhD, Principal Investigator — UMass Medical School; Anthony J. Windebank, MD, Principal Investigator — Mayo Clinic; Namita A. Goyal, MD, Principal Investigator — UC Irvine; Robert G. Miller, MD, Principal Investigator — California Pacific Medical Center (CPM) Research Institute; Robert Baloh, MD, Ph.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (6):
- United States (6):
  - University of California Irvine Alpha Stem Cell Clinic, Irvine, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant in Study BCT-002-US signed informed consent on 28 August 2017 The last participant visit took place on 29 September 2020. The study was conducted at 6 clinical sites in the USA. A total of 263 participants were screened for the study, and 196 participants (74.5% of participants screened) were randomly assigned (1:1) to treatment with either NurOwn or placebo.
Pre-assignment Details: The most common reasons that participants did not meet inclusion criteria were failure to meet the SVC inclusion criterion at the Screening Visit or the required pre-treatment decline in ALSFRSR total score at the randomization visit. From the ITT population, 3 participants in the NurOwn group and 4 participants in the placebo group discontinued prior to treatment.
Groups:
- NurOwn® (MSC-NTF Cells): NurOwn® (MSC-NTF): One course of treatment that includes three separate intrathecal injections of 100-125 x 10'6 cells every 8 weeks
  NurOwn® (MSC-NTF): Autologous, bone marrow-derived, mesenchymal stem cells secreting neurotrophic factors
  Bone marrow aspiration
- Placebo: One course of treatment that includes three separate intrathecal injections of Placebo every 8 weeks
  Placebo: liquid solution in syringe for injection
  Bone marrow aspiration
Period: Overall Study
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo
Started | 95 | 94
Completed | 71 | 73
Not Completed | 24 | 21
Not completed — Withdrawal by Subject | 12 | 14
Not completed — Death | 9 | 2
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Early Discontinuation | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographic characteristics were balanced between NurOwn and placebo treatment groups with no statistically significant differences at baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo | Total
Number analyzed (Participants) | 95 | 94 | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 94 | 189
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean | 48.1 (9.71) | 49.1 (8.38) | 48.6 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 35 | 62
  Male | 68 | 59 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 90 | 91 | 181
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 7 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 3 | 6
  White | 87 | 81 | 168
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 95 | 94 | 189
Baseline Amyotrophic Lateral Sclerosis Functional Rating ScaleScore [Mean (Standard Deviation); unit: units on a scale] — The ALSFRS-R is a quickly administered (10 minutes) ordinal, validated rating scale (ratings 0-4) used to determine participants' assessment of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Initial validity was established by documenting that in ALS patients, change in ALSFRS-R scores correlated with change in strength over time, as measured by quantitative neuromuscular strength testing, and with quality of life measures, and predicted survival. The total score of ALSFRS-R ranges from 0-48, with higher score being better.
  units on a scale | 30.3 (6.5) | 31.4 (6.1) | 30.9 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of NurOwn® Treated Participants With a ≥1.25 Points/Month Improvement in Post-treatment Slope vs. Pre-treatment Slope in ALSFRS-R Score at 28 Weeks Following the First Treatment as Compared to Placebo
Description: The ALSFRS-R is a quickly administered (10 minutes) ordinal, validated rating scale (ratings 0-4) used to determine participants' assessment of their capability and independence in 12 functional activities. All 12 activities are relevant in ALS. Initial validity was established by documenting that in ALS patients, change in ALSFRS-R scores correlated with change in strength over time, as measured by quantitative neuromuscular strength testing, and with quality of life measures, and predicted survival. The total score of ALSFRS-R ranges from 0-48, with higher score being better.
Time Frame: 28 weeks following the first intrathecal injection
Population: The modified intent-to-treat (mITT) population was defined as all participants who were randomized, treated and had at least three ALSFRS-R assessments: one pre-treatment assessments of ALSFRS-R prior to the baseline assessment, a baseline assessment and one post-treatment assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo
Number analyzed (Participants) | 95 | 94
Participants
  YES (%) | 31 | 26
  NO (%) | 64 | 68
Statistical Analysis 1: Comparison: NurOwn® (MSC-NTF Cells) vs Placebo; Test type: Superiority; p = 0.453, Chi-squared; Odds Ratio (OR) = 1.330, 95% CI 2-sided [0.632 to 2.798]

2. Secondary Outcome: Number of Participants Whose Disease Progression is Halted or Improved as Measured by a 100% or Greater Improvement in Post-treatment Slope vs. Pre-treatment Slope in ALSFRS-R Score of NurOwn® Treatment vs. Placebo
Description: as for outcome 1
Time Frame: 28 weeks following the first intrathecal injection
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo
Number analyzed (Participants) | 95 | 94
Participants
  YES (%) | 13 | 13
  NO (%) | 82 | 81
Statistical Analysis 1: Comparison: NurOwn® (MSC-NTF Cells) vs Placebo; Test type: Superiority; p = 0.997, Chi-squared; Odds Ratio (OR) = 0.998, 95% CI 2-sided [0.416 to 2.395]

3. Secondary Outcome: Score of NurOwn® (MSC-NTF Cells) Treated Patients vs. Placebo Treated Patients as Measured by Change From Baseline in ALSFRS-R Score at Week 28
Description: as for outcome 1
Time Frame: 28 weeks following the first intrathecal injection
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo
Number analyzed (Participants) | 95 | 94
score on a scale | -5.52 (0.670) | -5.88 (0.665)
Statistical Analysis 1: Comparison: NurOwn® (MSC-NTF Cells) vs Placebo; Test type: Superiority; p = 0.693, Mixed Models Analysis; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-1.47 to 2.20], Standard Error of Mean 0.926

4. Secondary Outcome: NurOwn® (MSC-NTF Cells) Treated Patients vs. Placebo Treated Patients as Measured by the Combined Assessment of Function and Survival at 28 Weeks
Description: The combined Assessment of Function and Survival (CAFS) is a composite endpoint based on (1) the change from baseline in ALS Functional Rating Scale-Revised (ALSFRS-R) score and (2) time to death.
  On the ALSFRS-R, 12 functions are rated on 5-point ordinal rating scales (from 0 to 4) with a total score range (minimum and maximum score) of 0-48 (sum of all 12 items). The higher the score the better functioning. For the survival endpoint, the longer time the better outcome.
  A patient's CAFS score represents a patient's rank in the study based on comparing the patient's outcome for both the change in ALSFRS-R and the time to death to all other patients in the study in a pairwise fashion. The ranked scores range from 001 to 189 (the number of subjects in the mITT population) with larger rank score numbers associated with a better outcome. The reported values are the mean rank scores in each group for the composite endpoint.
Time Frame: 28 weeks following the first intrathecal injection
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo
Number analyzed (Participants) | 95 | 94
score on a scale | 73.74 (5.210) | 72.21 (4.890)
Statistical Analysis 1: Comparison: NurOwn® (MSC-NTF Cells) vs Placebo; Test type: Superiority; p = 0.804, ANCOVA; Mean Difference (Final Values) = 1.53, 95% CI 2-sided [-10.65 to 13.72], Standard Error of Mean 6.176

ADVERSE EVENTS:
Time Frame: from the screening visit through the end of the study period (28 weeks after first treatment)
Description: AE means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Groups:
- NurOwn® (MSC-NTF Cells): NurOwn® (MSC-NTF): One course of treatment that includes three separate intrathecal injections of 100-125 x 10^6 cells every 8 weeks
  NurOwn® (MSC-NTF): Autologous, bone marrow-derived, mesenchymal stem cells secreting neurotrophic factors
  Bone marrow aspiration
Arm/Group | NurOwn® (MSC-NTF Cells) | Placebo
All-Cause Mortality (participants affected / at risk) | 10/95 | 4/94
Serious Adverse Events (participants affected / at risk) | 23/95 | 17/94
Other Adverse Events (participants affected / at risk) | 93/95 | 92/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NurOwn® (MSC-NTF Cells) (N=95) | Placebo (N=94)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 1 (1) | 2 (2)
Euthanasia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (3)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NurOwn® (MSC-NTF Cells) (N=95) | Placebo (N=94)
Procedural pain (Injury, poisoning and procedural complications) | 50 (145) | 34 (52)
Procedural headache (Injury, poisoning and procedural complications) | 31 (58) | 30 (51)
Fall (Injury, poisoning and procedural complications) | 28 (61) | 34 (76)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 22 (36) | 29 (48)
Post procedural complication (Injury, poisoning and procedural complications) | 16 (22) | 7 (10)
Contusion (Injury, poisoning and procedural complications) | 9 (9) | 9 (16)
Laceration (Injury, poisoning and procedural complications) | 7 (7) | 11 (12)
Postoperative fever (Injury, poisoning and procedural complications) | 7 (7) | 1 (2)
Limb injury (Injury, poisoning and procedural complications) | 6 (7) | 1 (2)
Procedural anxiety (Injury, poisoning and procedural complications) | 5 (7) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 5 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 42 (78) | 24 (33)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 (29) | 11 (15)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 (16) | 8 (9)
Coccydynia (Musculoskeletal and connective tissue disorders) | 11 (14) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 11 (15) | 12 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11) | 7 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (14) | 6 (6)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 7 (7) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (9) | 8 (8)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5)
Headache (Nervous system disorders) | 45 (85) | 32 (57)
Dizziness (Nervous system disorders) | 5 (6) | 5 (5)
Dysarthria (Nervous system disorders) | 2 (3) | 5 (6)
Balance disorder (Nervous system disorders) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 16 (20) | 18 (22)
Dysphagia (Gastrointestinal disorders) | 9 (9) | 5 (5)
Constipation (Gastrointestinal disorders) | 7 (7) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 7 (9)
Vomiting (Gastrointestinal disorders) | 3 (4) | 6 (6)
Pyrexia (General disorders) | 9 (10) | 9 (9)
Injection site pain (General disorders) | 8 (13) | 9 (10)
Chills (General disorders) | 2 (3) | 5 (5)
Fatigue (General disorders) | 0 (0) | 8 (8)
Nasopharyngitis (Infections and infestations) | 8 (8) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (8)
Anxiety (Psychiatric disorders) | 5 (5) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (5) | 3 (3)

LIMITATIONS AND CAVEATS:
This trial had a unique and atypical trial population that included more participants than anticipated with advanced ALS, who had a low ALSFRS-R score. As compared with recent large ALS clinical trials, this study population is an outlier, with a mean overall ALSFRS-R score at baseline lower than other studies, and this impacted the power of this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT03280056/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03280056/SAP_001.pdf